CLINICAL TRIAL: NCT04437550
Title: Effects of Exercise Intensity on Energy Intake, Appetite and Enjoyment in Overweight and Obese Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Marywood University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Marywood University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 801776
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity (Experimental)
  Interventions: Other: Exercise
- low-intensity (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — high intensity exercise = 15 x 60 s sprints at 85% velocity of VO2max (vVO2max) with 60 s walking at 20% vVO2max or moderate intensity exercise = walking at 60% vVO2max

SUMMARY:
Interval exercise involves short bouts of high intensity exercise interspersed with periods of lower intensity exercise. The benefit is that a shorter total duration of exercise may be required to achieve cardiovascular benefits similar to or even superior to traditional longer bouts of steady state endurance exercise. However how this type of exercise affects appetite and energy intake, particularly in overweight and obese females is not well known.

This study involves two trials of exercise, one at high intensity and one at low intensity, followed by a buffet lunch, in overweight and obese females.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Adult
3. apparently healthy
4. overweight or class I obese
5. eumenorrheic

Exclusion Criteria:

1. Diabetes
2. pregnancy
3. cardiovascular disease
4. greater than 1 hour of structured physical activity per week
5. thyroid disease
6. polycystic ovary disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 11 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in energy expenditure | immediately pre-breakfast, immediately pre-exercise, during exercise, and immediately post-exercise.
  caloric expenditure measured via indirect calorimetry
Change in energy intake | immediately post exercise
  measured via standardized lunch
Change in appetite | immediately pre-breakfast, immediately post-breakfast, immediately post-exercise and immediately pre-lunch
  measured via circulating hormones leptin and acylated ghrelin
Change in subjective hunger | baseline, immediately pre-exercise, immediately post-exercise, immediately pre-lunch, and immediately post-lunch
  via visual analogue scale 100 mm, higher scores indicate greater hunger

CONTACTS AND LOCATIONS:
Locations (1):
- Human Physiology Lab, Scranton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No